CLINICAL TRIAL: NCT05894499
Title: Cohort Survey on Shock and Anaphylaxis in Persons With Underlying Diseases Considered to Be at High Risk of Severe COVID-19 by Using Vaccination Information
Brief Title: Post-Marketing Safety Study in Japan of Shock and Anaphylaxis After Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) mRNA-1273 COVID-19 Vaccine in Persons in at High Risk of Severe COVID-19
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P915
Record Dates: First submitted 2023-06-05; First posted 2023-06-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants received 2 doses of mRNA-1273 vaccine approximately 4 weeks apart.

SUMMARY:
The goal of this study is to confirm the onset status of hypersensitivity reactions including shock and anaphylaxis observed after vaccination with this drug in persons with underlying diseases who are considered to have a high risk of severe exacerbation of COVID-19 and explore risk factors.

DETAILED DESCRIPTION:
Data collected from the JDMC Claims Database between May 2021 to November 2021.

ELIGIBILITY:
Inclusion Criteria:

* Participants registered to receive the mRNA-1273 vaccine in the Pep Up vaccination history Database
* Participants who have a history of vaccination with the mRNA-1273 vaccine in the Pep-Up vaccination history Database and the observation start date is at least 6 months prior to vaccination with the mRNA-1273 vaccine and have underlying diseases. Data period for confirmation of presence/absence of underlying disease is May 2021 to November 2021.

Exclusion Criteria:

* Underlying diseases that were determined undetectable by the pre-screening of JMDC
* Participants who did not consent to the questionnaire.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was selected from participants who were registered to receive the mRNA-1273 vaccine in the Pep Up vaccination history Database whose start date of observation in the claim database was within 6 months or more before vaccination with mRNA-1273 vaccine, and those who met the definition of underlying disease based on the claim data for 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 13309 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Hypersensitivity Reactions Including Shock and Anaphylaxis After Either Dose 1 and Dose 2 | Up to 2 days post vaccination after either the first or second vaccination

SECONDARY OUTCOMES:
Number of Participants With Hypersensitivity Reactions Including Shock and Anaphylaxis After Dose 1 | Up to 2 days post vaccination
Number of Participants With Hypersensitivity Reactions Including Shock and Anaphylaxis After Dose 2 | Up to 2 days post vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- CMIC Co., Ltd., Tokyo, Japan